CLINICAL TRIAL: NCT04233593
Title: Imaging the Neuroimmune Response to Lipopolysaccharide
Brief Title: Neuroimmune Response to Lipopolysaccharide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Kelly Cosgrove, Associate Professor, Yale University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1305011987
Record Dates: First submitted 2020-01-11; First posted 2020-01-18 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-06

CONDITIONS: Healthy
Keywords: PET TSPO Imaging; Microglia Activation/Proliferation; Lipopolysaccharide
MeSH Terms: interventions — Lipopolysaccharides

STUDY DESIGN:
Intervention Model Description: All subjects will complete one 120-minute [11C]PBR28 PET scan before and one scan 3-hours after lipopolysaccharide (LPS; 1.0ng/kg; IV) administration. A subset of subjects will complete a follow-up [11C]PBR28 PET scan 24+ hours after LPS.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LPS Challenge (Experimental): Subjects will undergo one 120-minute [11C]PBR28 PET scan before and one scan 3-hours after LPS administration (1.0ng/kg; IV).
  Interventions: Biological: Lipopolysaccharide
- LPS Follow-up (No Intervention): Subjects will undergo one 120-minute [11C]PBR28 PET scan 24+ hours after LPS.

INTERVENTIONS:
Biological: Lipopolysaccharide — Endotoxin E Coli
  Other Names: LPS
  Arms: LPS Challenge

SUMMARY:
In this study, healthy adult volunteers will undergo two positron emission tomography (PET) scans using the radiotracer [11C]PBR28 which binds to the 18kDa translocator protein (TSPO). Approximately 3 hours prior to the second [11C]PBR28 PET scan, lipopolysaccharide (LPS; endotoxin) will be administered to evoke a robust neuroimmune response. Subjects will also undergo behavioral and cognitive testing. Vital signs, subjective response, and peripheral cytokine levels will be assayed periodically throughout the experimental session.

Specific aims: Quantify the magnitude of neuroimmune response after a classical immune stimulus.

Secondary aims: Quantify changes in cognitive function after a classical immune stimulus.

Hypothesis: Individuals will exhibit a robust whole-brain neuroimmune response and impaired cognitive function after LPS.

ELIGIBILITY:
Inclusion Criteria:

1) Medically-healthy male and female subjects able to read/write English

Exclusion Criteria:

1. Subjects cannot meet DSM criteria for substance use disorder
2. Any psychiatric symptoms that could put the subject at risk by participating in the study including but not limited to suicidal or homicidal ideation, or suicide attempt within the last year
3. Pregnancy or breastfeeding;
4. Any current medical illness that could put the subjects at risk during the PET scan, or interfere with the PET or immunologic measures
5. Significant hepatocellular injury (as evidenced by AST or ALT levels greater than 5 times normal or a history of cirrhosis) will be exclusionary in order to reduce the risks associated with alcohol consumption
6. Subjects taking corticosteroids or other immunosuppressant drugs
7. Subjects with disorders affecting the brain, including but not limited to multiple sclerosis, history of stroke, brain tumors, intracranial bleeding, infection, or abscess.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2014-03-25 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Baseline TSPO Availability | Before LPS administration (baseline)
  Time-activity curves will be extracted from brain regions of interest and analyzed using multilinear analysis-1 (t*=30) incorporating the metabolite-corrected arterial input function to yield [11C]PBR28 total volumes of distribution (VT) across brain regions.

SECONDARY OUTCOMES:
Alcohol Dependence Scale (ADS) - questionnaire | baseline
  self-report questionnaire to determine severity of alcohol symptoms, 25 question multiple choice scale, range of 0-47 for a total score, with higher numbers indicating worse severity

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Cosgrove, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No